CLINICAL TRIAL: NCT01904981
Title: Comparison of Beta-blocker Versus Angiotensin Receptor Blocker for Suppression of Aneurysm Expansion in Patients With Small Abdominal Aortic Aneurysm and Hypertension (BASE Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0843
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2018-12

CONDITIONS: Small Abdominal Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atenolol (Experimental): Atenolol group
  Interventions: Drug: Beta-blocker-Atenolol 50mg, PO(peroral), Once daily
- Valsartan (Experimental): Valsartan group
  Interventions: Drug: Angiotensin receptor blocker-Valsartan 80mg, PO(peroral), Once daily

INTERVENTIONS:
Drug: Beta-blocker-Atenolol 50mg, PO(peroral), Once daily
  Arms: Atenolol
Drug: Angiotensin receptor blocker-Valsartan 80mg, PO(peroral), Once daily
  Arms: Valsartan

SUMMARY:
Various medical therapies have been proposed to prevent abdominal aortic aneurysm expansion. However, there have been very few randomized clinical trials to support use of any of these treatments. Several animal studies and observational reports suggest that ARBs can be useful in reducing abdominal aortic aneurysm (AAA) growth. However, so far, ARBs have not been evaluated in a randomized clinical trial. Therefore, the purpose of the study is to evaluate the effect of valsartan, an ARB, on annual growth rate in comparison with atenolol, a beta-blocker. Our hypothesis is that valsartan is superior to atenolol in the suppression of the aneurysm growth at 12 months. The BASE trial is designed as a investigator-initiated, multi-center, randomized controlled open-label trial. Patients with small AAA (aorta diameter <5cm) will be randomized 1:1 either to valsartan or to atenolol group. Randomization will be stratified by the AAA size (max. diameter >4 cm or ≤4 cm). Patients will receive either valsartan (daily dose 80 mg or more) or atenolol (daily dose 50 mg or more) for 12 months. A CT scan will measure the maximal diameter of AAA at baseline and 12 months. The annual growth of AAA will be compared between the valsartan and the atenolol group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20years
* Abdominal aortic aneurysm with maximal diameter less than 5cm
* Hypertension
* Patient with signed informed consent

Exclusion Criteria:

* Saccular type aneurysm, inflammatory aneurysm, or infected aneurysm
* Aortic dissection
* Planned surgery or endovascular therapy for abdominal aortic aneurysm within 1 year
* Previous aorta surgery or endovascular therapy
* Contraindications to Beta-blocker or ARB (allergic reactions, asthma, severe bradycardia, angioedema, hyperkalemia)
* Allergic reaction to contrast dye
* Known genetic aorta disease or autoimmune or connective tissue disease: Marfan syndrome, Shprintzen-Goldberg syndrome, Loeys-Dietz syndrome, Takayasu's arteritis, Behcet's disease
* Pregnancy
* Life expectation <1 year
* Renal failure (serum Cr >2.0 mg/dL)
* Liver disease (ALT or AST > 3 x upper limit) or liver cirrhosis (Child B or C)
* Malignancy requiring surgery or chemotherapy within 1 year after enrollment
* Status post transplantation or chronic inflammatory disease requiring immune suppressive drugs over 4 weeks

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Annual aneurysm growth of abdominal aortic aneurysm | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea